CLINICAL TRIAL: NCT05810974
Title: The Impact of Inorganic Nitrate-rich Beetroot Juice on Microvascular Blood Flow, Cognitive Function and Other Hemodynamic Outcomes in Postmenopausal Women
Brief Title: The Impact of Inorganic Nitrate-rich Beetroot Juice on Microvascular Blood Flow and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Charlotte E Mills, Lecturer, Principal investigator, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: -TBC-
Record Dates: First submitted 2023-02-08; First posted 2023-04-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-04

CONDITIONS: Post Menopausal
Keywords: Beetroot; NO; Nitrate; Microvascular function; Cognition
MeSH Terms: interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Concentrated beetroot juice (Active Comparator)
  Interventions: Dietary Supplement: Concentrated beetroot juice
- Nitrate depleted beetroot juice + potassium nitrate (KNO3) (Active Comparator)
  Interventions: Dietary Supplement: Nitrate depleted beetroot juice + potassium nitrate (KNO3)
- Nitrate-depleted beetroot juice (Placebo Comparator)
  Interventions: Dietary Supplement: Nitrate depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Concentrated beetroot juice — Subjects will consume 70ml shot (Beet-it Sport nitrate 400 shot, James White Drinks) and this drink contains 0.4g inorganic nitrate
  Arms: Concentrated beetroot juice
Dietary Supplement: Nitrate depleted beetroot juice + potassium nitrate (KNO3) — Nitrate-depleted beetroot juice (70ml) and 0.4g KNO3- will be mixed. (Same appearance and taste with Beet-it sport shot)
  Arms: Nitrate depleted beetroot juice + potassium nitrate (KNO3)
Dietary Supplement: Nitrate depleted beetroot juice — Subjects will consume 70ml of (Beet-it Placebo shot, James White Drinks). This drink is the same as the Beet-it Sport nitrate shot but has the nitrate removed.
  Arms: Nitrate-depleted beetroot juice

SUMMARY:
Cardiovascular disease (CVD) is one of the leading causes of mortality worldwide. Inorganic nitrate found in beetroot and green leafy vegetables has been demonstrated to reduce cardiovascular disease risk factors including reducing blood pressure and the stiffness of blood vessels by increasing levels of a compound called nitric oxide. Much of the research to date has focused on the large blood vessels, and little is known about the impact of inorganic nitrate on smaller blood vessels which could be related to cognitive function.

The majority of beneficial effects with inorganic nitrate have been observed within young healthy populations. However, it is known that after the menopause women are at an increased risk of cardiovascular disease and have reduced levels of nitric oxide in their body; this could also contribute to the cognitive decline also observed post-menopause. This trial will investigate the impact of inorganic nitrate from beetroot juice on the blood flow in small blood vessels and on cognitive function in postmenopausal women. The hypothesis of the study is that the nitrate in beetroot juice will increase circulating nitric oxide that will then increase blood flow in small blood vessels and improve cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy post-menopausal women (age over 45)
* Able to understand information sheet and willing to comply with the study protocol and able to give informed consent
* Not having menstrual period for 12 months

Exclusion Criteria:

* Blood pressure <90/60 or > 140/90 mmHg
* Medical history of myocardial infarction, angina, thrombosis, stroke, cancer, high cholesterol, liver, renal, respiratory or bowel diseases or diabetes or other endocrine disorder
* BMI>30
* Any tobacco and/or nicotine users (or quit within the last 6 months)
* Current use of antihypertensive medication
* Alcohol intake > 14 units/week
* Vigorous exercise > 3 times/ week
* Antihypertensive medication users
* People who have had hysterectomy
* Currently taking hormone replacement therapy or selective oestrogen receptor modulator

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline endothelial dependent microvascular function as laser Doppler imaging (LDI) with iontophoresis | At baseline (t= 0.5 hours) and t= 3 hours
  Measurements will be taken by LDI with iontophoresis of endothelium-dependent (acetylcholine (ACh))
Change from baseline endothelial independent microvascular function as laser Doppler imaging (LDI) with iontophoresis | At baseline (t= 0.5 hours) and t= 3 hours
  Measurements will be taken by LDI of endothelium-independent (sodium nitroprusside (SNP))
Change from baseline cognitive function. Domain: Episodic memory | At baseline (t= 0 hours) and t=2.5 hours
  -Rey Auditory Verbal Learning Test (RAVLT) task
  Cognitive domains will be assessed by using the Gorilla online research tools.
Change from baseline cognitive function. Domain: Executive function 1 | At baseline (t= 0 hours) and t=2.5 hours
  -Digit Span Task
Change from baseline cognitive function. Domain: Executive function 2 | At baseline (t= 0 hours) and t=2.5 hours
  -Stroop Task

SECONDARY OUTCOMES:
Change in blood pressure | [Time Frame: At baseline (t= 0 hours) and 15 minute intervals until t= 2.5 hours.]
  Systolic and Diastolic Blood pressure measurement by automated device

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No